CLINICAL TRIAL: NCT04779138
Title: Community Partnered Intervention to Increase COVID-19 Vaccine Uptake in Low Income Underresourced African Americans and Latinx Public Housing Residents
Brief Title: Increasing Vaccine Uptake in Underresourced Public Housing Areas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: vaccinehousing
Record Dates: First submitted 2021-02-27; First posted 2021-03-03 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-02

CONDITIONS: Coronavirus; Vaccine Refusal
MeSH Terms: conditions — Coronavirus Infections; Vaccination Refusal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Increasing Uptake of COVID-19 Vaccination (Experimental): This is a pre-experimental "one group pretest-posttest" design to increase COVID-19 vaccine uptake and completion among African American and Latinx public housing residents in South Los Angeles. The proposed intervention will employ (1) culturally sensitive, (2) theoretically based intervention that will be jointly delivered by our ACTIVATE triad leaders and our researchers. We will use the Information, Motivation, and Behavioral Skills (IMB) model and the Transtheoretical Model to implement the intervention.
  Interventions: Behavioral: Increasing Willingness and Uptake of COVID-19 Vaccination

INTERVENTIONS:
Behavioral: Increasing Willingness and Uptake of COVID-19 Vaccination — Provide/enhance knowledge, modify attitudes, motivate and provide skills and resources to reduce COVID-19 vaccine hesitancy and increase willingness and uptake in COVID-19 vaccination.

SUMMARY:
This proposal seeks to enhance uptake and completion of COVID-19 vaccination among African American and Latinx public housing residents in South Los Angeles. Given the multiple disparities experienced by public housing residents, the investigators will utilize a theoretically-based, multidisciplinary and culturally tailored intervention to provide education at multiple levels and implement innovate strategies to engage this population in the uptake of COVID-19 vaccination.

DETAILED DESCRIPTION:
One particular group, African American and Latinx public housing residents, are facing adverse effects related to worsening social determinants and health disparities. Utilizing a community-driven approach, the overall objective of this proposed study is to increase COVID-19 vaccine uptake and completion the impact of COVID-19 among African American and Latinx public housing residents. Guided by the Community Based Participatory Model, the Information, Motivation, and Behavioral Skills (IMB) and the Transtheoretical Model will be utilized to carry out this intervention. Through this innovative program, we will establish Academic-Community Team for Improving Vaccine Acceptability and Targeted Engagement (ACTIVATE) program, which will develop leadership triads of public housing resident leaders, nurse practitioner students, and public health students to carry out this multilevel intervention.

ELIGIBILITY:
Aim 2:

Inclusion Criteria:

* identify as Latinx or African American
* age 18 or older
* reside in one of the six collaborating public housing area
* Speak either English or Spanish

Exclusion Criteria:

* Not a resident at one of the collaborating public housing areas
* Does not self-identify as African American or Latinx
* Age 17 and younger
* Unable to speak either English or Spanish

Aim 3:

Inclusion Criteria:

* identify as Latinx or African American
* age 18 or older
* reside in one of the six collaborating public housing area
* Speak either English or Spanish
* Report vaccine hesitancy

Exclusion Criteria:

* Not a resident at one of the collaborating public housing areas
* Does not self-identify as African American or Latinx
* Age 17 and younger
* Unable to speak either English or Spanish
* Received all recommended vaccines for COVID-19
* No reporting of vaccine hesitancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of vaccination uptake for COVID-19, influenza, and pneumonia using Vaccination History Self Report | Intervention: 4 months; Follow-up Point: 3 months post-intervention
  1. By comparison of pre-, post- intervention, and 9- and 18-months follow-up data, we anticipate the following compared to baseline: a 40% change in completion of COVID-19 vaccination series

SECONDARY OUTCOMES:
Percentage of Participants Achieving Decreased Vaccine Hesitancy Levels of COVID-19 vaccine Using the NIH Toolbox Surveys on COVID-19 | Intervention: 4 months; Follow-up Point: 3 months post-intervention
  1. By comparison of pre-, post- intervention, and 3-months follow-up data, we anticipate the following compared to baseline: a 40% change in hesitancy toward COVID-19 vaccination.
Percentage of Participants Achieving Increased Level of Behavior Change toward COVID-19 Vaccination Using the NIH Toolbox Surveys on COVID-19 | Intervention: 4 months; Follow-up Point: 3 months post-intervention
  2. By comparison of pre-, post- intervention, and 3-months follow-up data, we anticipate the following compared to baseline: a 40% change in their behavior stage of change toward COVID-19 vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Cobb, Principal Investigator — Charles R. Drew University of Medicine & Science
Locations (1):
- Charles R. Drew University of Medicine & Science, Los Angeles, California, United States